CLINICAL TRIAL: NCT03270735
Title: A Multi-centre, Randomised, Double Blind, Placebo Controlled Clinical Study to Evaluate the Efficacy and Safety of Snake Venom Thrombin Injection in the Treatment of Moderate to Severe Hemoptysis
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of Hemocoagulase Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: Zhaoke Pharmaceutical (Hefei) Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-ZK-003
Record Dates: First submitted 2017-06-09; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-06

CONDITIONS: Hemoptysis
MeSH Terms: conditions — Hemoptysis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Snake venom thrombin
  Interventions: Drug: Snake venom thrombin (Treatment)
- Placebo (Placebo Comparator): Snake venom thrombin simulant
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Snake venom thrombin (Treatment) — Snake venom thrombin
  Other Names: Snake venom thrombin
  Arms: Treatment
Drug: Placebo — No snake venom thrombin
  Other Names: Snake venom thrombin simulant
  Arms: Placebo

SUMMARY:
This is a multi-centre, randomised, double blind, placebo controlled clinical study which is designed to evaluate the efficacy and safety of hemocoagulase in the treatment of moderate to severe hemoptysis.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years;
* Hemoptysis >=100 mL within 24 hours;
* Bronchiectasis diagnosed by chest high resolution CT;
* Patient, family or guardian is willing to sign the informed consent form.

Exclusion Criteria:

* With severe hepatic or renal insufficiency, ALT>3 ULN, creatinine clearance <30 mL/min or serum creatinine ≥200 µmol/L or ≥2.5 mg/dL;
* Uncontrollable hypertension (SBP>180mmHg or DBP>110mmHg) or hypotension shock (SBP<90 mmHg) at randomization;
* History of thrombosis, patients who have undergone thrombosis, or who have severe hematologic diseases;
* Patient with bleeding caused by DIC or vascular disease;
* Patient with coagulation dysfunction

  1. INR>2
  2. Patient with abnormal coagulation function or other bleeding disease (including clinical congenital bleeding disorders, such as von Willebrand disease or acquired hemophilia; hemorrhagic disease; and significant unexplained hemorrhagic disease)
  3. Platelet count <100×109 /L;
* known allergic to aspirin, clopidogrel, heparin, snake venom blood clotting enzyme, or any component in the study drug allergy or allergic constitution;
* Women who are pregnant or lactating and women of child-bearing agewho do not take reliable contraceptive measures;
* Patients who are or are planning to participate in other clinical trials during the study period;
* Within 72 hours before using the following products including Hemocoagulase For Injection (邦亭®), injection spearhead haemocoagulase (巴曲亭®), Haemocoagulase Agkistrodon for Injection (苏灵®), Hemocoagulase Atrox for Injection (立止血®), leaf pigment or other hemostatic agents;
* Life expectancy of less than 3 months;
* Any other patients who have been judged unfit to participate in this clinical study, including those who are unable or unwilling to comply with the protocol requirements;
* Patients who had participated in other clinical studies within three months prior to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
AEs and SAEs | 7 days
  The incidence of AEs and SAEs

SECONDARY OUTCOMES:
Effective rate of treating hemoptysis | 72 hours
  Effective rate of treating hemoptysis 72 hours after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, China